CLINICAL TRIAL: NCT00757211
Title: A Population Based Study of Genetic Predisposition and Gene-Environment Interactions in Breast Cancer in East Anglia
Brief Title: Study of Genes and Environment in Patients With Breast Cancer in the East Anglia Region of the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000598878; MREC-SEARCH-BREAST; MREC-07/MRE05/17
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at genetic susceptibility to cancer and interactions between genes and the environment in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain epidemiological information and biological material on a population-based series of breast cancer cases.
* To establish whether polymorphisms in putative cancer predisposition genes are associated with an increased risk of breast cancer by comparing the frequency of alterations in breast cancer patients with the corresponding frequency in controls.
* To define the proportion of breast cancer incidence attributable to mutations in such genes.
* To examine the interactions between genetic and nongenetic risk factors.
* To evaluate the relationship between pathological and clinical characteristics of breast cancers and germline genotype.

OUTLINE: This is a multicenter study.

Patients complete an epidemiological questionnaire that covers standard known breast cancer risk factors including reproductive history, oral contraceptive use, hormone replacement therapy use, family history, and alcohol consumption. The questionnaire will also request identifying information on the patient's first-degree relatives.

Blood samples are collected from patients. DNA is extracted from these blood samples, from samples collected from cancer-free control participants in MREC-SEARCH-CONTROL, and from additional controls through the European Prospective Investigation of Cancer (EPIC) study (a population-based study of diet and health based in Norfolk, East Anglia). DNA samples are analyzed for polymorphisms of low penetrance cancer susceptibility genes.

In addition to the breast cancer patients recruited for this study, patients with malignant melanoma and lymphoma, colorectal, ovarian, prostate, colorectal, bladder, kidney, pancreatic, and esophageal cancer, and brain tumors are recruited for the following related clinical trials: MREC-SEARCH-COLORECTAL, MREC-SEARCH-OVARIAN, MREC-SEARCH-PROSTATE, MREC-SEARCH-ENDOMETRIAL, and MREC-SEARCH-CANCER.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer within the past 5 years
* Identified through the East Anglian Cancer Registry in the East Anglia region of the United Kingdom
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Identified by the patient's general practitioner as fit to contact for this study
* No serious mental illness or retardation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Acquisition of epidemiological information and biological material
Investigation of whether polymorphisms in putative cancer predisposition genes are associated with an increased risk of breast cancer
Proportion of breast cancer incidence attributable to mutations in such genes
Examination of the interactions between genetic and nongenetic risk factors
Evaluation of the relationship between pathological and clinical characteristics of breast cancers and germline genotype

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pharoah, MD, Study Chair — Cancer Research UK
Locations (1):
- University of Cambridge Cancer Research UK, Cambridge, England, United Kingdom